CLINICAL TRIAL: NCT01886300
Title: A Multicenter, Prospective, Observational, Non-Interventional Cohort Study Evaluating Sustained Response in Subjects With HBeAg Positive Chronic Hepatitis B Receiving Therapy With Pegasys (Peginterferon Alfa-2a) in Vietnam
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) in Patients With HBeAg-Positive Chronic Hepatitis B in Vietnam
Status: Terminated | Type: Observational
Why Stopped: Due to out-of-date design and non-compliance.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27807
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multicenter, observational study will evaluate the sustained response in patients with HBeAg positive chronic hepatitis B who are treated with Pegasys according to standard of care and in line with the current local labeling in routine clinical practice in Vietnam. Eligible patients will be followed for the duration of their treatment and for up to 2 years thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* HBeAg-positive serologically proven chronic hepatitis B with or without cirrhosis
* Elevated serum ALT > ULN (upper limit of normal) but </= 10 x ULN
* Patients with no contra-indications to Pegasys therapy as detailed in the label
* Written informed consent where local regulations allow or require it

Exclusion Criteria:

* Patients should not receive concomitant therapy with telbivudine
* Co-infection with hepatitis A, hepatitis B or HIV
* Pregnant or breastfeeding women
* Patients with depression/mental diseases
* Neutrophil at baseline > 90.000/mm3
* Abnormal T4 or TSH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HBeAg-positive chronic hepatitis B treated with Pegasys
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Vietnam (3):
  - Hanoi
  - Ho Chi Minh City
  - Hochiminh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 335 participants planned to be enrolled in the study, only 16 participants were enrolled. The trial was conducted at 8 centers in Vietnam.
Groups:
- Peginterferon Alfa-2a: Participants with hepatitis B envelope antigen (HBeAg) positive chronic hepatitis B who received peginterferon alfa-2a [Pegasys] were included.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a
Started | 16
Completed | 0
Not Completed | 16
Not completed — Trial terminated by sponsor | 16

BASELINE CHARACTERISTICS:
Groups:
- Peginterferon Alfa-2a: Participants with HBeAg positive chronic hepatitis B who received peginterferon alfa-2a were included.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — As the sample size requirement for the study was not met, the study was terminated; no data for any of the participants was collected.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — As the sample size requirement for the study was not met, the study was terminated; no data for any of the participants was collected.
  Male | NA — As the sample size requirement for the study was not met, the study was terminated; no data for any of the participants was collected.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of Hepatitis B Virus Deoxyribonucleic Acid To <2,000 IU/mL at 6 Months After End of Treatment
Description: A participant was considered to have achieved suppression of Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) to <2,000 International Units Per Milliliter (IU/mL) if the HBV DNA measurement is lower than 2,000 IU/mL.
Time Frame: 6 months
Population: As the sample size requirement for the study was not met, the study was terminated; no data for any of the participants was collected.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Participants Who Become Hepatitis B Envelope Antigen-Negative and Anti-HBe-Positive During Treatment and at 6 and 12 Months After End of Treatment
Description: HBeAg is a protein from the Hepatitis B virus that circulates in infected blood when the virus is actively replicating. The presence of HBeAg suggests that the participant is infectious and is able to spread the virus to other people. HBeAg-negative hepatitis B is a form of the virus that does not cause infected cells to secrete HBeAg. Participant can be infected with the HBeAg-negative form of the virus from the beginning, or the viral mutation can emerge later in the course of infection in participant initially infected with the HBeAg-positive form of the virus.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Suppression of Hepatitis B Virus Deoxyribonucleic Acid To <2,000 IU/mL During the Observation Period
Description: A participant was considered to have achieved suppression of HBV DNA to <2,000 IU/mL if the HBV DNA measurement is lower than 2,000 IU/mL.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Loss of Hepatitis B Envelope Antigen During the Observation Period
Description: Loss of HBeAg is defined as the absence of HBeAg. A participant was considered to have achieved HBeAg loss if the HBeAg measurement was reported as (a) 'NEGATIVE' or (b) a quantitative result was lower than the reported lower detection limit.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With Hepatitis B Envelope Antigen Seroconversion and Hepatitis B Virus Deoxyribonucleic Acid Suppression (<2,000 IU/mL) During the Observation Period
Description: HBeAg seroconversion is defined as the absence of HBeAg and the presence of antibody to hepatitis B antigen (anti-HBe) . A participant was considered to have achieved suppression of HBV DNA to <2,000 IU/mL if the HBV DNA measurement is lower than 2,000 IU/mL.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Who Become Hepatitis B Envelope Antigen Negative During the Observation Period
Description: as for outcome 2
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Normalization of Serum Alanine Transaminase
Description: Normalization of alanine transaminase (ALT) values means that ALT values out of the normal range returned to within the normal range.
Time Frame: Up to 24 months
Population: as for outcome 1
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Incidence of Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product
Time Frame: Up to 24 months
Population: Participants present at the time of assessment were used for analysis.
Measure: Number; unit: Number of participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 16
Number of participants | 9

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a (N=16)
Increasing HBV DNA (Investigations) | 1
Weight loss (Investigations) | 2
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Blurred Vision (Eye disorders) | 1
Flu symptom (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Transaminase Flare (Hepatobiliary disorders) | 1
Libido (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the sponsor's intellectual property rights.